CLINICAL TRIAL: NCT03207100
Title: Clinical Study of the Safety and Efficacy of Analgesia-first Minimal Sedation as an Early Antihypertensive Treatment for Spontaneous Intracerebral Hemorrhage
Brief Title: Analgesia-first Minimal Sedation for Spontaneous Intracerebral Hemorrhage Early Antihypertensive Treatment
Acronym: ASSICHH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Yang (Other Government)
Collaborators: Xuanwu Hospital, Beijing (Other); Qilu Hospital of Shandong University (Other); First Affiliated Hospital of Kunming Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Second Affiliated Hospital of Third Military Medical University (Other); Henan Provincial People's Hospital (Other); The Second Hospital University of South China (Other); Shenzhen Second People's Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Department of Biostatistics, Southern Medical University (Unknown); LanZhou University (Other); The First Affiliated Hospital of HuNan University of Medicine (Unknown); Guangdong 999 Brain Hospital (Other); Maoming People's Hospital (Other); The Fifth Affiliated Hospital of Southern Medical University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Hong Yang, Doctor of Medicine (M.D.)；Associate Senior Doctor, The Third Affiliated Hospital of Southern Medical University
Organization: The Third Affiliated Hospital of Southern Medical University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201704004
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Early Systolic Blood Pressure Control Rate; Hematoma Growth; Blood Pressure Variability; Healthcare Worker Satisfaction; Duration of ICU Treatment and Mechanical Ventilation
Keywords: Intracerebral hemorrhage; Early antihypertensive treatment; Analgesia-first; Sedation
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: Subjects are grouped into the analgesia-first minimal sedation group (experimental group) or antihypertensive drug treatment group (control group) using the central randomization system upon enrollment. Antihypertensive intervention is performed on the subjects in accordance to the protocol of each group.
Who Masked: Participant
Masking Description: This study uses a single-blinded design in which only the investigators and not the subjects know the method of intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analgesia-first minimal sedation group (Experimental): Using analgesia-first minimal sedation strategy to implement antihypertensive therapy.
  Interventions: Combination Product: Analgesia-first minimal sedation
- Antihypertensive drug treatment group (Active Comparator): Using routine antihypertensive drugs to implement antihypertensive therapy.
  Interventions: Combination Product: Antihypertensive treatment

INTERVENTIONS:
Combination Product: Analgesia-first minimal sedation — Remifentanil will be administered by IV infusion and maintained at a dose of 0.025 μg/kg/min in non-mechanically ventilated patients and a dose of 0.05 μg/kg/min in mechanically ventilated patients. BP will be measured after 10 min of continuous infusion.If systolic BP is still ≥ 140 mmHg, then dexmedetomidine will be applied using an infusion pump at a dose of 0.2 μg/kg/h. BP will be measured again after 15 min of continuous infusion of dexmedetomidine. If systolic BP is still ≥ 140 mmHg, the dose of dexmedetomidine can be increased 0.1 μg/kg/h to the maximum of 0.6 μg/kg/h.If the maximum dose of dexmedetomidine does not lower blood pressure, use routine blood pressure reduction programs in each center to reduce blood pressure to the target range. Mechanically ventilated patients will be given a rapid remifentanil (0.5 μg/kg) infusion to reduce procedure-related pain.
  Arms: Analgesia-first minimal sedation group
Combination Product: Antihypertensive treatment — Routine antihypertensive treatment will be performed in accordance with the protocol of each respective research center. Urapidil, nicardipine, and labetalol will be used in this group. Urapidil will be used as follows: a slow IV injection of 10-15 mg and then IV pumping for maintenance at an initial rate of 2 mg/min, adjusted according to BP to a maximum of 9 mg/min. Nicardipine will be used as follows: IV pumping at 0.5μg/kg/min adjusted according to BP to a maximum of 6μg/kg/min. Labetalol will be used as follows: IV infusion for maintenance at 1-4 mg/min until the aim is reached.The mechanically ventilated patients in the control group will be administered a rapid physiological saline infusion as a controlled pretreatment.
  Arms: Antihypertensive drug treatment group

SUMMARY:
This study evaluates safety and efficacy of analgesia-first minimal sedation as an early antihypertensive treatment for spontaneous intracerebral hemorrhage. The analgesia-first minimal sedation strategy relies on the remifentanil-mediated alleviation of pain-induced stress response and the antisympathetic activity of dexmedetomidine to restore the elevated blood pressure to normal level in patients with spontaneous intracerebral hemorrhage. This strategy allows rapid stabilization of blood pressure, and its use as a pre-treatment for patients on mechanical ventilation prior to painful procedures reduces blood pressure variability and thereby results in etiologic treatment. It is more effective in blood pressure control than conventional symptomatic antihypertensive treatment, reduces the incidence of early hematoma expansion and improves prognosis, ,lowers healthcare workers workload, increases patient adherence, and improves healthcare worker satisfaction.

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage (ICH) is hemorrhage in the brain parenchyma caused by non-traumatic spontaneous rupture of cerebral artery, arteriole, vein and capillary in adults. ICH is a common problem, with subarachnoid hemorrhage. About 90% ICH patients have increased blood pressure (BP) that usually occurs immediately after disease onset. BP elevation in the acute phase of ICH is associated with poor prognosis, and its mechanism of action includes the local increase of initial hemorrhage, early hematoma expansion at hemorrhagic sites, the increased risk of early recurrent hemorrhage, serious cerebral edema, and recurrent stroke, this affects the most within the few hours following the onset of the disease. The current American Heart Association guidelines recommended early antihypertensive treatment and suggested that rapid decrease of BP to 140 mmHg is safe in ICH patients with no obvious antihypertensive contraindications. However, the significant differences between large studies conducted in recent years have led to great controversy on the effect of early antihypertensive treatment in acute ICH and disease prognosis. A meta-analysis of early antihypertensive treatment for ICH showed that differences in early BP control rate and BP increase variability are also the major causes of inconsistency between these studies. There is currently no consensus on the best antihypertensive regimen as it is difficult to reach the optimal BP level timely. Some studies have shown that stress response, pain, ICP increase and pre-onset BP elevation are factors that cause acute BP increase in ICH patients. In particular, restlessness, sleep deprivation, and stress due to intolerable pain can lead to dramatic BP and intracranial pressure (ICP) increases, further lead to secondary intracerebral hematoma expansion and subsequently cause neurologic degeneration and cerebral tissue damage. Therefore, the primary principles of ICH acute BP increase treatment are to keep quiet, restore BP to normal level, stably reduce BP, decrease BP variability, lower the chance of recurrent hemorrhage, and thereby improve long-term prognosis. Traditional antihypertensive treatment can only resolve the issue of BP elevation but not the root cause of disease. Analgesia and sedation is a critical component of and a global consensus in the clinical management of ICH patients. Remifentanil is a fentanyl μ-type opioid receptor agonist with strong and fast-acting analgesic effects, does not induce ICP elevation and can alleviate pain induced by sputum aspiration, body turning and back clapping in severe patients. A randomized trial on patients with craniocerebral injury has indicated that a remifentanil-based sedation strategy can significantly reduce the amount of sedative used and shorten the time of mechanical ventilation without affecting the functional assessment of the nervous system. Dexmedetomidine is an α2-adrenergic agonist that inhibits sympathetic activity by activating the pre-synaptic α2-receptor in the locus coeruleus, which in turn reduces norepinephrine release, that only slightly affects consciousness and breathing and helps patients with craniocerebral injury stay conscious while under sedation, allowing real-time functional assessment of the nervous system. Therefore, the research group developed a treatment strategy in which sufficient analgesia is applied in combination with a minimal sedation program as an effective and safe early an- tihypertensive treatment.We hypothesize that applying sufficient analgesia in combination with a minimal sedation program will involve the use of remifentanil for pain relief and dexmedetomidine for antisympathetic activity to restore elevated BP to normal levels in patients with spontaneous ICH, and we further hypothesize that this strategy will be more effective than conventional symptomatic antihypertensive treatment for controlling BP.

ELIGIBILITY:
Inclusion Criteria:

1. Definitive diagnosis of ICH-induced acute brain injury by CT;
2. Systolic BP ≥150 mmHg for at least twice;
3. >18 years old;
4. Feasible for emergency antihypertensive treatment and real-time BP monitoring;
5. Disease onset is within 24h;
6. ICU or stroke unit admission within 24h.

Exclusion Criteria:

1. Subject has contraindications for emergency intensified antihypertensive treatment;
2. Intracranial hemorrhage secondary to intracranial tumor, recent trauma, cerebral infarction and thrombolytic therapy;
3. History of ischemic stroke within 30 days before disease onset;
4. Clinical or imaging examination reveals an expected high mortality in subject within the next 24h;
5. Presence of dementia or significant post-stroke disability;
6. Coagulation disorder caused by drugs or hematologic diseases;
7. Allergy to opioids;
8. Interference test result, assessment and follow-up of comorbidity;
9. Presence of sinus arrest, borderline rhythm, grade II and above atrioventricular block and malignant arrhythmia;
10. Individual is pregnant or lactating;
11. Currently participating in other drug studies or clinical trials;
12. Subject or guardian is unwilling to provide his/her informed consent form, or subject is highly unable to persist with the study and follow-up;
13. Subject's participation in the study will increase his/her study-related risk, and other reasons that make the subject unsuitable for the study as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2021-02-14 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Systolic BP control rate at 1h post-treatment initiation | 1h post-treatment initiation
  The number of patients who systolic BP decreased to <140 mmHg at 1h post-treatment initiation compared to the total number of each group.

SECONDARY OUTCOMES:
Hematoma growth at 24 h | 24h of treatment
  Head CT re-examination is required for the subjects after 24h of treatment.Hematoma expansion is defined as V2-V1≥12.5 cm³ or (V2-V1)/V1>33% (V1 and V2 represent the hematoma volume in the two CT scans, respectively).
BP variability | Up to 7 days
  BPs are also recorded every hour from hour 2 to 24 post-treatment, and monitored on d2-d7 of treatment of recorded every 6h daily (4 times per day); BP Coefficient of Variation (CV) = (standard deviation of BP/mean of systolic BP).
Neurologic function | Up to 7 days
  Assessed once every morning using the National Institutes of Health Stroke Scale (NIHSS), Glasgow Coma Scale scores (GCS), Richmond Agitation-Sedation Scale (RASS), Nonverbal Adult Pain Assessment Scale (NVPS), Reaction Level Scale (RLS).
Duration of ICU treatment and mechanical ventilation | Up to 7 days
  Duration of ICU treatment and mechanical ventilation
Healthcare worker satisfaction | 7 day or discharge from ICU (if patients discharge from ICU in 7 days)
  Questionnaire is designed based on the Copenhagen Psychosocial Questionnaire, with a parameter for self-assessed workload.
cerebral tissue oxygenation index (TOI) | Up to 7 days and around sputum aspiration
  Assess changes in the TOI after sputum aspiration in mechanical ventilation patients
28-day mortality and disability rate | 28 days
  Using a binary indicator of the patient's death or dependency at 28 days, with dependency being defined by a score of 3 to 5 on the modified Rankin Score (mRS)
90-day mortality and disability rate | 90 days
  Using a binary indicator of the patient's death or dependency at 90 days, with dependency being defined by a score of 3 to 5 on the modified Rankin Score (mRS)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jin Chen, Study Chair — Xuanwu Hospital, Beijing; Hong Yang, Dr, Study Chair — The Third Affiliated Hospital of Southern Medical University
Locations (17):
- China (17):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Xinqiao Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong 999 Brain Hospital, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - MaoMing People's Hospital, Maoming, Guangdong
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The Fifth Affiliated Hospital Sun-yet sen University, Zhuhai, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Second Hospital University of South China, Hengyang, Hunan
  - The First Affiliated Hospital of HuNan University of Medicine, Huaihua, Hunan
  - Qilu Hospital of Shandong University, Qingdao, Shandong
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kuming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qureshi AI, Tuhrim S, Broderick JP, Batjer HH, Hondo H, Hanley DF. Spontaneous intracerebral hemorrhage. N Engl J Med. 2001 May 10;344(19):1450-60. doi: 10.1056/NEJM200105103441907. No abstract available. PMID 11346811
- [Background] Chen ST, Chen SD, Hsu CY, Hogan EL. Progression of hypertensive intracerebral hemorrhage. Neurology. 1989 Nov;39(11):1509-14. doi: 10.1212/wnl.39.11.1509. PMID 2812332
- [Background] Broderick JP, Brott TG, Tomsick T, Barsan W, Spilker J. Ultra-early evaluation of intracerebral hemorrhage. J Neurosurg. 1990 Feb;72(2):195-9. doi: 10.3171/jns.1990.72.2.0195. PMID 2295917
- [Background] Arakawa S, Saku Y, Ibayashi S, Nagao T, Fujishima M. Blood pressure control and recurrence of hypertensive brain hemorrhage. Stroke. 1998 Sep;29(9):1806-9. doi: 10.1161/01.str.29.9.1806. PMID 9731599
- [Background] van Swieten JC, Koudstaal PJ, Visser MC, Schouten HJ, van Gijn J. Interobserver agreement for the assessment of handicap in stroke patients. Stroke. 1988 May;19(5):604-7. doi: 10.1161/01.str.19.5.604. PMID 3363593
- [Background] Koskinen LO, Olivecrona M, Grande PO. Severe traumatic brain injury management and clinical outcome using the Lund concept. Neuroscience. 2014 Dec 26;283:245-55. doi: 10.1016/j.neuroscience.2014.06.039. Epub 2014 Jun 25. PMID 24973658
- [Background] Stocchetti N, Pagan F, Calappi E, Canavesi K, Beretta L, Citerio G, Cormio M, Colombo A. Inaccurate early assessment of neurological severity in head injury. J Neurotrauma. 2004 Sep;21(9):1131-40. doi: 10.1089/neu.2004.21.1131. PMID 15453984
- [Background] Oddo M, Crippa IA, Mehta S, Menon D, Payen JF, Taccone FS, Citerio G. Optimizing sedation in patients with acute brain injury. Crit Care. 2016 May 5;20(1):128. doi: 10.1186/s13054-016-1294-5. PMID 27145814
- [Background] Broderick JP, Brott TG, Duldner JE, Tomsick T, Huster G. Volume of intracerebral hemorrhage. A powerful and easy-to-use predictor of 30-day mortality. Stroke. 1993 Jul;24(7):987-93. doi: 10.1161/01.str.24.7.987. PMID 8322400
- [Background] Kazui S, Naritomi H, Yamamoto H, Sawada T, Yamaguchi T. Enlargement of spontaneous intracerebral hemorrhage. Incidence and time course. Stroke. 1996 Oct;27(10):1783-7. doi: 10.1161/01.str.27.10.1783. PMID 8841330
- [Background] Kasner SE. Clinical interpretation and use of stroke scales. Lancet Neurol. 2006 Jul;5(7):603-12. doi: 10.1016/S1474-4422(06)70495-1. PMID 16781990
- [Background] Teasdale G, Maas A, Lecky F, Manley G, Stocchetti N, Murray G. The Glasgow Coma Scale at 40 years: standing the test of time. Lancet Neurol. 2014 Aug;13(8):844-54. doi: 10.1016/S1474-4422(14)70120-6. PMID 25030516
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the Intensive Care Unit: executive summary. Am J Health Syst Pharm. 2013 Jan 1;70(1):53-8. doi: 10.1093/ajhp/70.1.53. PMID 23261901
- [Background] Stalhammar D, Starmark JE, Holmgren E, Eriksson N, Nordstrom CH, Fedders O, Rosander B. Assessment of responsiveness in acute cerebral disorders. A multicentre study on the reaction level scale (RLS 85). Acta Neurochir (Wien). 1988;90(3-4):73-80. doi: 10.1007/BF01560558. PMID 3354366
- [Background] Pejtersen JH, Kristensen TS, Borg V, Bjorner JB. The second version of the Copenhagen Psychosocial Questionnaire. Scand J Public Health. 2010 Feb;38(3 Suppl):8-24. doi: 10.1177/1403494809349858. PMID 21172767
- [Result] Wallace JD, Levy LL. Blood pressure after stroke. JAMA. 1981 Nov 13;246(19):2177-80. PMID 7289008
- [Result] Harper G, Castleden CM, Potter JF. Factors affecting changes in blood pressure after acute stroke. Stroke. 1994 Sep;25(9):1726-9. doi: 10.1161/01.str.25.9.1726. PMID 8073450
- [Result] Ong TZ, Raymond AA. Risk factors for stroke and predictors of one-month mortality. Singapore Med J. 2002 Oct;43(10):517-21. PMID 12587706
- [Result] Becker KJ, Baxter AB, Bybee HM, Tirschwell DL, Abouelsaad T, Cohen WA. Extravasation of radiographic contrast is an independent predictor of death in primary intracerebral hemorrhage. Stroke. 1999 Oct;30(10):2025-32. doi: 10.1161/01.str.30.10.2025. PMID 10512902
- [Result] Mayer SA, Sacco RL, Shi T, Mohr JP. Neurologic deterioration in noncomatose patients with supratentorial intracerebral hemorrhage. Neurology. 1994 Aug;44(8):1379-84. doi: 10.1212/wnl.44.8.1379. PMID 8058133
- [Result] Zhou JF, Wang JY, Luo YE, Chen HH. Influence of hypertension, lipometabolism disorders, obesity and other lifestyles on spontaneous intracerebral hemorrhage. Biomed Environ Sci. 2003 Sep;16(3):295-303. PMID 14631835
- [Result] Kazui S, Minematsu K, Yamamoto H, Sawada T, Yamaguchi T. Predisposing factors to enlargement of spontaneous intracerebral hematoma. Stroke. 1997 Dec;28(12):2370-5. doi: 10.1161/01.str.28.12.2370. PMID 9412616
- [Result] Gebel JM Jr, Jauch EC, Brott TG, Khoury J, Sauerbeck L, Salisbury S, Spilker J, Tomsick TA, Duldner J, Broderick JP. Natural history of perihematomal edema in patients with hyperacute spontaneous intracerebral hemorrhage. Stroke. 2002 Nov;33(11):2631-5. doi: 10.1161/01.str.0000035284.12699.84. PMID 12411653
- [Result] Carhuapoma JR, Hanley DF, Banerjee M, Beauchamp NJ. Brain edema after human cerebral hemorrhage: a magnetic resonance imaging volumetric analysis. J Neurosurg Anesthesiol. 2003 Jul;15(3):230-3. doi: 10.1097/00008506-200307000-00010. PMID 12826970
- [Result] Anderson CS, Heeley E, Huang Y, Wang J, Stapf C, Delcourt C, Lindley R, Robinson T, Lavados P, Neal B, Hata J, Arima H, Parsons M, Li Y, Wang J, Heritier S, Li Q, Woodward M, Simes RJ, Davis SM, Chalmers J; INTERACT2 Investigators. Rapid blood-pressure lowering in patients with acute intracerebral hemorrhage. N Engl J Med. 2013 Jun 20;368(25):2355-65. doi: 10.1056/NEJMoa1214609. Epub 2013 May 29. PMID 23713578
- [Result] Delcourt C, Huang Y, Wang J, Heeley E, Lindley R, Stapf C, Tzourio C, Arima H, Parsons M, Sun J, Neal B, Chalmers J, Anderson C; INTERACT2 Investigators. The second (main) phase of an open, randomised, multicentre study to investigate the effectiveness of an intensive blood pressure reduction in acute cerebral haemorrhage trial (INTERACT2). Int J Stroke. 2010 Apr;5(2):110-6. doi: 10.1111/j.1747-4949.2010.00415.x. PMID 20446945
- [Result] Qureshi AI, Mohammad YM, Yahia AM, Suarez JI, Siddiqui AM, Kirmani JF, Suri MF, Kolb J, Zaidat OO. A prospective multicenter study to evaluate the feasibility and safety of aggressive antihypertensive treatment in patients with acute intracerebral hemorrhage. J Intensive Care Med. 2005 Jan-Feb;20(1):34-42. doi: 10.1177/0885066604271619. PMID 15665258
- [Result] Terayama Y, Tanahashi N, Fukuuchi Y, Gotoh F. Prognostic value of admission blood pressure in patients with intracerebral hemorrhage. Keio Cooperative Stroke Study. Stroke. 1997 Jun;28(6):1185-8. doi: 10.1161/01.str.28.6.1185. PMID 9183348
- [Result] Anderson CS, Huang Y, Wang JG, Arima H, Neal B, Peng B, Heeley E, Skulina C, Parsons MW, Kim JS, Tao QL, Li YC, Jiang JD, Tai LW, Zhang JL, Xu E, Cheng Y, Heritier S, Morgenstern LB, Chalmers J; INTERACT Investigators. Intensive blood pressure reduction in acute cerebral haemorrhage trial (INTERACT): a randomised pilot trial. Lancet Neurol. 2008 May;7(5):391-9. doi: 10.1016/S1474-4422(08)70069-3. Epub 2008 Apr 7. PMID 18396107
- [Result] Manning L, Hirakawa Y, Arima H, Wang X, Chalmers J, Wang J, Lindley R, Heeley E, Delcourt C, Neal B, Lavados P, Davis SM, Tzourio C, Huang Y, Stapf C, Woodward M, Rothwell PM, Robinson TG, Anderson CS; INTERACT2 investigators. Blood pressure variability and outcome after acute intracerebral haemorrhage: a post-hoc analysis of INTERACT2, a randomised controlled trial. Lancet Neurol. 2014 Apr;13(4):364-73. doi: 10.1016/S1474-4422(14)70018-3. Epub 2014 Feb 13. PMID 24530176
- [Result] Kate MP, Hansen MB, Mouridsen K, Ostergaard L, Choi V, Gould BE, McCourt R, Hill MD, Demchuk AM, Coutts SB, Dowlatshahi D, Emery DJ, Buck BH, Butcher KS; ICHADAPT Investigators. Blood pressure reduction does not reduce perihematoma oxygenation: a CT perfusion study. J Cereb Blood Flow Metab. 2014 Jan;34(1):81-6. doi: 10.1038/jcbfm.2013.164. Epub 2013 Sep 18. PMID 24045403
- [Result] Boulouis G, Morotti A, Goldstein JN, Charidimou A. Intensive blood pressure lowering in patients with acute intracerebral haemorrhage: clinical outcomes and haemorrhage expansion. Systematic review and meta-analysis of randomised trials. J Neurol Neurosurg Psychiatry. 2017 Apr;88(4):339-345. doi: 10.1136/jnnp-2016-315346. Epub 2017 Feb 18. PMID 28214798
- [Result] Egawa S, Hifumi T, Kawakita K, Okauchi M, Shindo A, Kawanishi M, Tamiya T, Kuroda Y. Impact of neurointensivist-managed intensive care unit implementation on patient outcomes after aneurysmal subarachnoid hemorrhage. J Crit Care. 2016 Apr;32:52-5. doi: 10.1016/j.jcrc.2015.11.008. Epub 2015 Dec 2. PMID 26703419
- [Result] Rodriguez-Luna D, Pineiro S, Rubiera M, Ribo M, Coscojuela P, Pagola J, Flores A, Muchada M, Ibarra B, Meler P, Sanjuan E, Hernandez-Guillamon M, Alvarez-Sabin J, Montaner J, Molina CA. Impact of blood pressure changes and course on hematoma growth in acute intracerebral hemorrhage. Eur J Neurol. 2013 Sep;20(9):1277-83. doi: 10.1111/ene.12180. Epub 2013 May 5. PMID 23647568
- [Result] Tanaka E, Koga M, Kobayashi J, Kario K, Kamiyama K, Furui E, Shiokawa Y, Hasegawa Y, Okuda S, Todo K, Kimura K, Okada Y, Okata T, Arihiro S, Sato S, Yamagami H, Nagatsuka K, Minematsu K, Toyoda K. Blood pressure variability on antihypertensive therapy in acute intracerebral hemorrhage: the Stroke Acute Management with Urgent Risk-factor Assessment and Improvement-intracerebral hemorrhage study. Stroke. 2014 Aug;45(8):2275-9. doi: 10.1161/STROKEAHA.114.005420. Epub 2014 Jun 26. PMID 24968929
- [Result] Li M, Zhang Y, Wu KS, Hu YH. Assessment of the effect of continuous sedation with mechanical ventilation on adrenal insufficiency in patients with traumatic brain injury. J Investig Med. 2016 Mar;64(3):752-8. doi: 10.1136/jim-2015-000012. Epub 2016 Feb 10. PMID 26912007
- [Result] Balestreri M, Czosnyka M, Chatfield DA, Steiner LA, Schmidt EA, Smielewski P, Matta B, Pickard JD. Predictive value of Glasgow Coma Scale after brain trauma: change in trend over the past ten years. J Neurol Neurosurg Psychiatry. 2004 Jan;75(1):161-2. PMID 14707332
- [Result] Engelhard K, Reeker W, Kochs E, Werner C. Effect of remifentanil on intracranial pressure and cerebral blood flow velocity in patients with head trauma. Acta Anaesthesiol Scand. 2004 Apr;48(4):396-9. doi: 10.1111/j.0001-5172.2004.00348.x. PMID 15025597
- [Result] Yokota H, Yokoyama K, Noguchi H, Nishioka T, Umegaki O, Komatsu H, Sakaki T. Post-operative dexmedetomidine-based sedation after uneventful intracranial surgery for unruptured cerebral aneurysm: comparison with propofol-based sedation. Neurocrit Care. 2011 Apr;14(2):182-7. doi: 10.1007/s12028-010-9485-4. PMID 21174172
- [Result] Grof TM, Bledsoe KA. Evaluating the use of dexmedetomidine in neurocritical care patients. Neurocrit Care. 2010 Jun;12(3):356-61. doi: 10.1007/s12028-008-9156-x. PMID 20217277
- [Result] Kothari RU, Brott T, Broderick JP, Barsan WG, Sauerbeck LR, Zuccarello M, Khoury J. The ABCs of measuring intracerebral hemorrhage volumes. Stroke. 1996 Aug;27(8):1304-5. doi: 10.1161/01.str.27.8.1304. PMID 8711791
- [Result] Topolovec-Vranic J, Canzian S, Innis J, Pollmann-Mudryj MA, McFarlan AW, Baker AJ. Patient satisfaction and documentation of pain assessments and management after implementing the adult nonverbal pain scale. Am J Crit Care. 2010 Jul;19(4):345-54; quiz 355. doi: 10.4037/ajcc2010247. PMID 20595216
- [Derived] Dong R, Li F, Xu Y, Chen P, Maegele M, Yang H, Chen W. Safety and efficacy of applying sufficient analgesia combined with a minimal sedation program as an early antihypertensive treatment for spontaneous intracerebral hemorrhage: a randomized controlled trial. Trials. 2018 Nov 6;19(1):607. doi: 10.1186/s13063-018-2943-6. PMID 30400977